CLINICAL TRIAL: NCT04332055
Title: Measuring the Effect of an ePRO-based Clinical Decision Support System in Knee- and Hip Replacement Surgery
Brief Title: RCT Measuring the Effect of the ERVIN Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2015-141-ERVIN
Record Dates: First submitted 2020-03-06; First posted 2020-04-02 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-03

CONDITIONS: Decision Making, Shared; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip; Osteoarthritis, Knee; Osteoarthritis, Hip; Artificial Intelligence
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to the two intervention arms using a randomised block design stratified by age, Oxford Hip- or Knee Score at baseline and location of disability. Age and Oxford scores are subdivided into suitable categories20. Randomization will be done using REDCap electronic data capture21. Block sizes will be random with possible volumes of four and eight patients. Patients will be randomised after completion of the survey questions at the ePRO kiosk. Information regarding randomisation will be typed in separate REDCap module by the designated helper, after which a randomisation key is automatically generated, which can then be extracted by the designated helper, but blinded from the patient.
Who Masked: Participant
Masking Description: Patients are blinded from the randomisation, and blinding of the consulting surgeon is not possible since the intervention is an interface add-on to the conventional treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERVIN PLUS (Experimental): The doctor and the patient will have access to the ERVIN generated data
  Interventions: Other: ERVIN
- ERVIN MINUS (No Intervention): The doctor and the patient will not have access to the ERVIN generated data

INTERVENTIONS:
Other: ERVIN — ERVIN is state of the art for IT systems, which uses artificial intelligence (AI) and real-time patient-specific PRO data to support patients and doctors in clinical decision-making. The system is designed for surgical OA treatment of knee and hip replacement, and can be used to predict outcome scores for the actual choice OA patients face in the patient trajectory; to choose surgery or not.
  Arms: ERVIN PLUS

SUMMARY:
The randomised clinical trial investigates the effect of using a clinical decision support system (CDSS) aiming to provide the patients and surgeons with greater transparency concerning the obtainable changes in function and health related quality of life (HRQoL) when patients are to decide if they should undergo hip- or knee replacement surgery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) affects 20 % of the adult population in Denmark, and the economic burden to society is estimated to DKK 4.6 billion per year1,2. Symptoms related to evolving OA can usually be effectively managed, and treatment may slow the progression of the disease, however, approximately 10,000 and 8,000 hip and knee replacements, respectively, are performed each year in Denmark due to end-stage OA3-5.

The Danish clinical guidelines for the treatment of OA are compliant with international guidelines and recommend non-pharmacological and complementary pharmacological treatment as first-line treatment modalities3. When non-surgical treatment options become insufficient to relieve pain and improve function, referral to an orthopaedic surgeon for evaluation of whether the patient is eligible for surgery is advised. However, the guidelines do not provide clear guidance on which non-pharmacological treatment(s) or when surgery will be most beneficial for the individual patient, and consequently under- or over-utilisation of healthcare services may occur 3,6 Furthermore, matching patient's expectations with the achievable changes in function level after surgery can be challenging, which might be a contributor to the 20 % proportion of orthopaedic patients that are unsatisfied7,8. It highlights the importance of an enhanced basis for shared decision-making between surgeon and patient, as-well-as bringing focus on each patient's wishes and needs, as these are individual and thus might not be representative of the general population.

Patient-centred care acknowledges the importance of individual values and preferences and empowers patients to take an active part in decisions concerning their health and treatment pathway9. It moves beyond the paternalistic approach to treatment, substituting in its place a partnership-like relation between patient and clinician9,10.

Patient reported outcomes (PRO) have been suggested as a means to improve patient involvement and patient value through a shift in the perception of what constitute "good outcomes", and PRO has on several occasions been shown to be important predictors of clinical outcomes11-13. PRO measures are available for most clinical areas, but implementing a more patient-centred health-care system through PRO is still challenged by i.a. information asymmetry, and lack of aligning expectations12,14.

Denmark has a long tradition of collecting patient-specific data in the health care sector. The challenge today is that the knowledge embedded in these patient-specific health-care data is not utilized to its full potential, neither within nor between the primary and the secondary health care sectors, and, currently, there is a lack of knowledge on how to incorporate data and ePRO (electronic Patient Reported Outcome) to support patients in clinical decision-making.

ERVIN is state of the art for IT systems, which uses artificial intelligence (AI) and real-time patient-specific PRO data to support patients and doctors in clinical decision-making. The system is designed for surgical OA treatment of knee and hip replacement, and can be used to predict outcome scores for the actual choice OA patients face in the patient trajectory; to choose surgery or not.

The clinical and health economic rationale for this study is three-folded: one, to explore if the use of real-time, and predicted ePRO in clinical decision-making impacts patients health; two, to investigate if the use of ERVIN enhances shared decision-making in clinical practice, and third, to investigate if the use of ERVIN is cost-effective.

This study aims to establish the health-related effect and cost-effectiveness of using ERVIN in clinical consultation when the OA patient is referred from the general practitioner to orthopaedic clinic to decide if the patient should have a total hip- or knee replacement.

The increased focus and endorsement of patient-centred care and increased patient involvement in clinical decisions in the Danish health care system is a result of political decisions. The health-related consequences of practising patient centred-care, where patients are more empowered to make decisions are unknown. Furthermore, there is a lack of knowledge of how, and under which conditions, CDDS solutions, like ERVIN, create value in health15,16.

Objective The main objective of this randomised controlled trial is to investigate the health related effects of using ERVIN as a CDSS during consultations, measured by the delta value in Oxford Hip Score (OHS) and Oxford Knee Score (OKS) pre- and post-treatment modalities. Secondary outcomes include investigations of cost-effectiveness and the degree of shared decision-making.

Hypothesis The hypothesis is that the application of ERVIN in consultations, compared with the conventional approach in surgical decision-making concerning hip- or knee replacement, do not lead to any change in OHS or OKS between baseline and at 1-year follow-up.

Methods

Trial design The implementation of ERVIN to enhance patient-centeredness is based on a shift in the government policy for the Danish Health Care system. The new strategy requires increased use of digital solutions in health care and improvement of patient involvement in decisions making17,18. However, the impact on patients' health, when patient involvement is increased by the use of a digital solution like ERVIN is unknown, and for that reason, a non-inferiority design is chosen in the trial.

The trial is a single centre, randomised, controlled trial, which includes two parallel groups. The intervention- and the control group will both have the conventional approach available during the consultation, which includes: A 25-minute consultation in which the surgeon evaluates the need/no need for surgery based on; the patients' subjective description of pains and disabilities, and general health. If available, a description of the aforementioned evaluation criteria from the referring general practitioner will be included in addition to the orthopaedic surgeons' evaluation of relevant x-rays and possible MRI or CT-scans and a physical examination.

The intervention group will have the results from ERVIN as an interface with a graphical presentation of real-time and predicted outcome scores and risk scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred from a general practitioner in the North Denmark Region to the orthopaedic clinic at Aalborg University Hospital
* Patients with painful OA in hip- or knee joint.

Exclusion Criteria:

* Patients unable to answer the questions in danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Oxford Hip Score | 1 year
  The OHS is a short 12-item PRO questionnaire, which is specifically designed and developed to assess the primary outcome in randomised controlled trials with patients undergoing hip or knee replacement surgery. The questionnaires are reproducible, validated and sensitive to clinically important changes24. The primary outcome measure is the delta value in OHS, or OKS measured at baseline, defined as the first consultation in the clinic, and at 1-year follow-up.
Oxford Knee Score | 1 year
  The OKS is a short 12-item PRO questionnaire, which is specifically designed and developed to assess the primary outcome in randomised controlled trials with patients undergoing hip or knee replacement surgery. The questionnaires are reproducible, validated and sensitive to clinically important changes24. The primary outcome measure is the delta value in OHS, or OKS measured at baseline, defined as the first consultation in the clinic, and at 1-year follow-up.

SECONDARY OUTCOMES:
HRQoL | 1 year
  as measures of effect in the economic evaluations. HRQoL is measured by the 15 item questionnaire; EQ-5D-3L
SDM | 2 hours
  SDM is measured by two 9-item Shared Decision Making Questionnaires; SDM-Q-9 (patient version), and SDM-Q-Doc (physician version)

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Kastrup, MSc, Principal Investigator — DCHI
Locations (1):
- Nanna Kastrup, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kastrup N, Bjerregaard HH, Laursen M, Valentin JB, Johnsen SP, Jensen CE. An AI-based patient-specific clinical decision support system for OA patients choosing surgery or not: study protocol for a single-centre, parallel-group, non-inferiority randomised controlled trial. Trials. 2023 Jan 12;24(1):24. doi: 10.1186/s13063-022-07039-5. PMID 36635747